CLINICAL TRIAL: NCT00830245
Title: A Study to Assess the Efficacy of Erlotinib for Leptomeningeal Carcinomatosis in EGFR Mutation Positive Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual rate
Sponsor: Clinical Research Center for Solid Tumor, Korea (Other)
Collaborators: Seoul National University Hospital (Other); Korean Cancer Study Group (Other)
Responsible Party: Dae Seog Heo/Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRCST-L-0005
Record Dates: First submitted 2009-01-24; First posted 2009-01-27 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Leptomeningeal Carcinomatosis; Non-small Cell Lung Cancer
Keywords: EGFR mutation; Erlotinib; Lung cancer; leptomeningeal carcinomatosis in EGFR mutation positive non-small cell lung cancer
MeSH Terms: conditions — Meningeal Carcinomatosis; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Erlotinib (Experimental): Erlotinib 150mg/day (if no negative conversion --> increment to 250mg/day)
  Interventions: Drug: Erlotinib

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150mg/day

SUMMARY:
To assess the efficacy and safety of erlotinib for non-small cell lung cancer patients with leptomeningeal carcinomatosis

ELIGIBILITY:
Inclusion Criteria:

1. Age >18
2. Histologically or pathologically proven non-small cell lung cancer (NSCLC)
3. Leptomeningeal carcinomatosis confirmed by CSF cytology
4. A patients with EGFR mutation (including exon 19 deletion, L858R)
5. ECOG performance status 0-3
6. Expected life time more than at least 4 weeks
7. A patients who signed the informed consent prior to the participation in the study
8. Chemotherapy-naïve patient is eligible
9. Previous EGFR TKI is allowed if this drug was not specifically used for CNS metastases

Exclusion Criteria:

1. A pregnant or lactating patient
2. A patient of childbearing potential without being tested for pregnancy at baseline or with a positive test. (A postmenopausal woman with the amenorrhea period of at least 12 months or longer is considered to have non-childbearing potential.)
3. A man or woman of childbearing potential without the willingness to use a contraceptive measures during the study
4. A patient with history of another malignant disease within past 3 years, except curatively treated basal cell carcinoma of the skin, cervical carcinoma in situ, and early gastric cancer
5. A patient with active interstitial lung disease, except simple lymphangitic lung metastasis
6. A patient with history of allergic reaction to gefitinib or erlotinib
7. The following laboratory test results:

   * Number of absolute neutrophils counts (ANC) < 1.0ⅹ109/L
   * Number of platelets < 50 ⅹ109/L
   * AST, ALT > 2.5 ⅹupper limit of normal
   * Total bilirubin > 1.5 ⅹupper limit of normal
   * Serum creatinine > 1.5 ⅹupper limit of normal
8. A patient with serious disease as followings

   * Uncontrolled cardiac arrhythmia
   * History of myocardial infarction within 6 months prior to the initiation of study
   * Neurological or psychiatric disorder including dementia or uncontrolled seizure
9. A patient who refused to sign the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Overall survival | 1 year

SECONDARY OUTCOMES:
Cytology negative conversion rate | 1 month, 2 months, 3 months, 4 months
Neurologic symptom improvement | 1 month, 2 months, 3 months, 4 months
Response rate (extra-cranial disease) | 2 months, 4 months
Response rate (brain) | 2 months, 4 months
Quality of life | 1 month, 2 months, 3 months, 4 months
Toxicities | 1 month, 2 months, 3 months, 4 months
Prognostic factors | N-A

CONTACTS AND LOCATIONS:
Locations (1):
- Dae Seog Heo, Seoul, South Korea